CLINICAL TRIAL: NCT01647555
Title: Prospective Study About the Association of Radiotherapy and Cetuximab in the Treatment of Epidermoid Cancers, Locally Advanced, of the Head and Neck.
Brief Title: Radiotherapy in Association With Cetuximab in Patients Treated for an Epidermoid Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: ESPACE
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Epidermoid Head and Neck Cancer
Keywords: Cetuximab; radiotherapy; epidermoid head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient with epidermoid cancer: receiving Cetuximab and radiotherapy
  Interventions: Drug: Cetuximab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — First cycle: 400 mg/m2 Next cycles: 250 mg/m2
Radiation: Radiotherapy — Curative dose: 66 to 70 Gy

SUMMARY:
This study evaluates the skin toxicities in patients with epidermoid cancer, treated by Radiotherapy in association with Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Epidermoid head and neck carcinoma locally advanced
* Indication of Cetuximab and radiotherapy
* Karnofsky >= 60
* Patients participating to another compatible study could be included after consultation with the study director Patients could be beforehand treated for an other ORL cancer

The radiotherapy will be delivered for curative aim (minimal dose 66 Gy)

Exclusion Criteria:

* other histology
* Metastatic disease
* Recurrent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with epidermoid head and neck cancer locally advanced
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2006-11; Primary Completion 2012-05 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Skin toxicities | until week 38
  according to NCI-CTCAE version 3.0

SECONDARY OUTCOMES:
Healthcare and evolution of skin toxicities | until week 38
  Treatment of skin toxicities, according to sponsor advices.
Quality of life | baseline, week 4, month 6
  Questionnaire QLQ-C30
tumoral efficacy | 6 months after treatment
  According to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Eric LARTIGAU, MD PhD, Study Director — Oscar Lambret Center
Locations (7):
- France (7):
  - Clinique du Parc, Croix
  - Centre Leonard de Vinci, Douai
  - Centre Bourgogne, Lille
  - Centre Oscar Lambret, Lille
  - Centre Galilée, Lille
  - Centre Gray, Maubeuge
  - Centre Joliot Curie, Saint Martin Les Boulogne